CLINICAL TRIAL: NCT06441955
Title: Covid-19 Long Haul Syndrome: Undiagnosed Disorder Post Covid-19 Alternative Treatment Study.
Brief Title: Covid-19 Long Haul Preventative and Health Promotion Care Clinical Trial Acceleration Program.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Well- Konnect Healthcare Services and Research Firm (Network)
Collaborators: All of Us Research Program at the National Institute of Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: aou-rw-c6288c3f
Record Dates: First submitted 2024-06-02; First posted 2024-06-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: COVID-19, Long Haul
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — nirmatrelvir and ritonavir drug combination; 2019-nCoV Vaccine mRNA-1273; Psychotherapy; DNA, Recombinant

STUDY DESIGN:
Intervention Model Description: A parallel study is a type of clinical study in which two or more groups of participants receive different interventions. Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial. Assignment to a group usually is randomized. Study participants are only exposed to the treatment that is assigned to the particular study arm they are enrolled in.
  For example, a two-arm parallel assignment involves two groups of participants. One group receives drug A, and the other group receives drug B. So during the trial, participants in one group receive drug A "in parallel" to participants in the other group, who receive drug B.
Masking Description: Covid-19 Long Haul Preventative and Health Promotion Care Clinical Trial Acceleration Program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Moderna COVID-19 Vaccine (Active Comparator): Unvaccinated individuals: Two doses of Moderna COVID-19 Vaccine (2023-2024 Formula) are administered. The second dose is administered 1 month after the first. Moderna COVID-19 Vaccine to include the 2023-2024 formula. The Moderna COVID-19 Vaccine (2023-2024 Formula) includes a monovalent (single) component that corresponds to the Omicron variant XBB.1.5 of SARS-CoV-2. The Moderna COVID-19 Vaccine (2023-2024 Formula) is authorized for all doses administered to individuals 6 months through 11 years of age to prevent COVID-19. The Moderna COVID-19 Vaccine, Bivalent is no longer authorized for use in the United States. Moderna COVID-19 Vaccine is a suspension for injection. A single dose is 0.25 mL. (3) History of a severe allergic reaction (e.g., anaphylaxis) to any component of Moderna COVID-19 Vaccine or following a previous dose of a Moderna COVID-19 vaccine.
  Interventions: Drug: Ritonavir-Boosted Nirmatrelvir (Paxlovid); Diagnostic Test: Physiological Evaluation; Biological: Moderna COVID-19 Vaccine; Behavioral: Biopsychological; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling); Genetic: Genetic (including gene transfer, stem cell and recombinant DNA); Combination Product: Multidisciplinary approach
- Ritonavir-Boosted Nirmatrelvir (Paxlovid) (Active Comparator): The COVID-19 Treatment Guidelines Panel (the Panel) recommends using nirmatrelvir 300 mg with ritonavir 100 mg (Paxlovid) orally (PO) twice daily for 5 days in nonhospitalized adults with mild to moderate COVID-19 who are at high risk of disease progression (). Treatment should be initiated as soon as possible and within 5 days of symptom onset. Ritonavir-boosted nirmatrelvir is available through an FDA EUA for the treatment of mild to moderate COVID-19 in nonhospitalized adolescents aged 12 to 17 years and weighing ≥40 kg.4 For recommendations on using ritonavir-boosted nirmatrelvir in nonhospitalized children with COVID-19.
  Interventions: Drug: Ritonavir-Boosted Nirmatrelvir (Paxlovid); Diagnostic Test: Physiological Evaluation; Biological: Moderna COVID-19 Vaccine; Behavioral: Biopsychological; Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling); Genetic: Genetic (including gene transfer, stem cell and recombinant DNA); Combination Product: Multidisciplinary approach

INTERVENTIONS:
Drug: Ritonavir-Boosted Nirmatrelvir (Paxlovid) — Participant Selection and Baseline Data Collection: 6 months
  * Longitudinal Observation and Intervention Implementation: 24 months
  * Data Analysis and Findings Dissemination: 6 months Evaluate methodological advantages and limitations of an international pharmacosurveillance system based on electronic health records (EHRs). Adverse outcome; Electronic health record; Health informatics; Medication adherence; Pharmacoepidemiology; Pharmacosurveillance; Risk assessment.
  Other Names: Phramacotherapies
Diagnostic Test: Physiological Evaluation — Common Medical laboratory work-up, Cancer screening test, Biomarkers, tissue biopsy, blood specimen, diagnostic imagining, Sensitivity and Specificity, HIV PCR, Viral load ( antigen), CD4- T cell count, while implementation of social mediators of prevention, promotion studies and conceptual models and quality of care.
  Other Names: Immunologic Evaluation
Biological: Moderna COVID-19 Vaccine — Single dose, 0.25 mL If previously vaccinated, ≥2 months after receipt of the last previous dose of COVID-19 vaccine
Behavioral: Biopsychological — Diagnosis of developmental milestones is considered a missing element in care measurement or a determining factor in disease signs and symptoms in chronic care management. Cognitive mapping, variations of survey, assessments, cancer counseling, leading to the realization that adherence requires a whole-person approach to delivering high-quality and cost-effective care. the project aims to offer opportunities to individuals from diverse backgrounds, including those underrepresented in biomedical research, in an inclusive environment in which all trainees can contribute. The proposed training activities are designed to improve the research skills of the participants and encourage them to pursue further training and careers in biomedical and/or social/behavioral research.
Behavioral: Behavioral (e.g., Psychotherapy, Lifestyle Counseling) — Diagnosis of developmental milestones is considered a missing element in care measurement or a determining factor in disease signs and symptoms in chronic care management. Cognitive mapping, variations of survey, assessments, cancer counseling, leading to the realization that adherence requires a whole-person approach to delivering high-quality and cost-effective care. the project aims to offer opportunities to individuals from diverse backgrounds, including those underrepresented in biomedical research, in an inclusive environment in which all trainees can contribute. The proposed training activities are designed to improve the research skills of the participants and encourage them to pursue further training and careers in biomedical and/or social/behavioral research.
  Other Names: Biopsychological
Genetic: Genetic (including gene transfer, stem cell and recombinant DNA) — Full genome sequencing, complete genome sequencing, or entire genome sequencing, is the process of determining the entirety, or nearly the entirety, of the DNA sequence of an organism's genome at a single time to address the intersection of genomics and health disparities, recognizing that genetic variations can contribute to health disparities in several ways. Understanding these genetic contributions to health disparities is crucial for developing targeted interventions and personalized healthcare strategies that can help address these disparities. genetics, epidemiology, public health, and social sciences, the study aims to shed light on the complex interplay between genomics and health equity. To evaluate cellular errors and the effects of myocardial DNA, you may need to consider tests such as DNA sequence.
  Other Names: Whole Genome Sequence
Combination Product: Multidisciplinary approach — The aim of utilizes psychology-applied science and science in nursing frameworks to address health disparities and promote health and wellness across the health span to improve patient population outcomes, evaluate cost-effectiveness, and patient health literacy competencies. The experimental framework of a compilation of the bio-psychosocial model, Eric Erickson developmental stages, AI/AML, and cognitive learning theories address system decision making factors, for sound decision making and behavioral change cognitive behavioral therapies protocol segmentation demographic and urban areas affected by social-economic access to healthcare and related ethical stance of United States healthcare policy developmental outlines. Biology plays a role in the content of development stages, and the great debate of nurture vs. nature sets the foundation for addressing the psychosocial approach to healthcare integration as an applied science model for strengthening primary services and improving

SUMMARY:
Investigators are conducting a study on alternative treatments for patients who have received an current or previous positive COVID-19 diagnosis with mild-serve symptoms or undiagnosable condition after testing positive for severe acute COVID-19 infection and are experiencing long-haul symptoms. The symptoms of long COVID can include extreme tiredness (fatigue), shortness of breath, memory and concentration issues (brain fog), heart palpitations, dizziness, joint pain, muscle aches, cough, headaches, anxiety, and depression.

It's important to note that there are various other symptoms that individuals can experience after a COVID-19 infection, such as loss of smell, chest pain or tightness, difficulty sleeping (insomnia), pins and needles, depression, anxiety, tinnitus, earaches, nausea, diarrhea, stomach aches, loss of appetite, cough, headaches, sore throat, and changes to the sense of smell or taste.

To be included in the study, participants must have had symptoms for more than 4 weeks. The goal of the study is to measure biomarkers, identify new ones through clinical trials, and individualize and optimize treatment plans, which may or may not include COVID-19 post-market antivirals, vaccines, and medical care.

It's essential to conduct thorough clinical trials to understand the long-term effects of COVID-19 and to develop personalized treatment plans for individuals experiencing long-haul symptoms.

DETAILED DESCRIPTION:
Investigators are planning a comprehensive study to understand and address the long-term effects of COVID-19. Investigators aim to recruit 25 to 100 participants who have tested positive or clinically diagnosed with COVID-19, regardless of whether they have received treatment with COVID-19 post-market antivirals, vaccines, or medical care. The study will involve conducting intake eligibility assessments and providing available treatments for COVID-19 to address the core morbidities associated with long-haul COVID-19.

Investigators plans also includes collecting data from diverse participants to define seven biomarker categories and create a prognosis indicator for COVID-19 symptoms using precision medicine methods. The focus will be on neurological and respiratory symptoms affecting quality of life, with a special emphasis on women and men who are prone to developing Post COVID-19 long-haul syndrome. Additionally, participants have outlined a diversity plan to ensure representation from a wide range of demographics.

It's clear that you are dedicated to addressing the impact of long-haul COVID-19 and are taking a comprehensive approach to understand and treat the persistent symptoms experienced by individuals post-COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of Men, Women, and Minorities
* Participants must be at least 18 years old.
* Participants must have a positive COVID-19 diagnosis or clinical diagnosis of COVID-19
* Participants must have experienced persistent symptoms after recovering from the acute phase of the illness.
* Participants must be willing to provide informed consent to participate in the study.
* Participants must be able to communicate effectively in English or have a translator available.
* Participants must be able to attend follow-up appointments as required by the study protocol.
* Participants must not have any medical conditions or take any medications that could interfere with the study results.

Exclusion Criteria:

* >18 years of age
* Medical History of Myocarditis
* Medical History of Pericarditis
* Medical History of Severe renal impairment (eGFR <30 mL/min).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence | - Participant Selection and Baseline Data Collection: 36 months - Longitudinal Observation and Intervention Implementation: 24 months - Data Analysis and Findings Dissemination: 36 months
  Well-Konnect Biopsychosoical Framework and assessment tool (WKBF tool) compared to the APA biopsychological assessment.
  Health literacy surveillance care program evaluation tool aims to lay the groundwork for a more inclusive and equitable approach to leveraging genomic data and interventions to improve health outcomes for all individuals.

SECONDARY OUTCOMES:
Pharmaco surveillance | - Participant Selection and Baseline Data Collection: 36 months - Longitudinal Observation and Intervention Implementation: 24 months - Data Analysis and Findings Dissemination: 36 months
  Evaluate methodological advantages and limitations of an international pharmacosurveillance system based on electronic health records (EHRs). Adverse outcome; Electronic health record; Health informatics; Medication adherence; Pharmacoepidemiology; Pharmacosurveillance; Risk assessment.

OTHER OUTCOMES:
Patient Engagement | - Participant Selection and Baseline Data Collection: 36 months - Longitudinal Observation and Intervention Implementation: 24 months - Data Analysis and Findings Dissemination: 36 months
  The research will delve into the impact of epigenetic factors on health outcomes, particularly in marginalized communities. By examining genomics and health equity, the study seeks to identify disparities in the prevalence and treatment of epigenetic conditions among different population groups. The goal is to develop targeted interventions and metrics to improve health outcomes and access to genomic interventions for all individuals, irrespective of their background or socioeconomic status.

CONTACTS AND LOCATIONS:
Overall Officials: Kawana J Williams, Ph.D., Principal Investigator — The National Institute of Health All of Us Research Program At Well-Konnect Healthcare Services and Research Center
Locations (1):
- NIH Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
No participant count of 1 to 20 can be published or distributed directly (a count of 0 is permitted); and No data or statistics can be reported that allow a participant count of 1 to 20 to be derived from other reported cells or information, including in text, tables, or figures.
Supporting Information: CSR, Analytic Code
Time Frame: 10 years
Access Criteria: Authorization for access to the registered and controlled data tiers will be user based, rather than project-based. Authorized users will receive a "data passport." A data passport is required for access to the registered and controlled data tiers and to set up workspaces to carry out research projects .
  As one of the first steps in initiating an All of Us registered and controlled tier project and setting up a workspace, users will be required to submit a description of their project. These descriptions will be made public and searchable for auditing purposes to facilitate public engagement.